CLINICAL TRIAL: NCT02385201
Title: Multi-Center, Prospective, Clinical Trial of the Senza™ Spinal Cord Stimulation (SCS) System in the Treatment of Chronic Upper Limb and Neck Pain
Brief Title: Clinical Trial of the Senza™ SCS System in the Treatment of Chronic Upper Limb and Neck Pain
Acronym: SENZA-ULN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nevro Corp (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA2014 US
Record Dates: First submitted 2015-03-03; First posted 2015-03-11 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Neck Pain; Chronic Pain
MeSH Terms: conditions — Neck Pain; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Senza (Experimental): Subjects with chronic, intractable pain of the upper limbs and/or neck will be implanted with a Senza Spinal Cord Stimulation (SCS) system designed to deliver electrical stimulation to the spinal cord.
  Interventions: Device: Senza

INTERVENTIONS:
Device: Senza — Spinal Cord Stimulation

SUMMARY:
This is a prospective, multi-center feasibility study of effectiveness and safety of the Senza System in subjects with chronic, intractable pain of the upper limbs and/or neck. Data at follow-up visits will be compared to Baseline data collected at the beginning of the study.

DETAILED DESCRIPTION:
Study subjects will be identified from the pool of candidates for SCS therapy affiliated with, or referred to, the clinical sites. Subjects will participate in this investigational plan that includes entry criteria evaluation, Baseline assessments, trial stimulation phase, and post-trial assessment. Subjects with a successful Trial Phase will receive a permanent implant of an Implantable Pulse Generator (IPG) and leads, and undergo 12 months of stimulation delivery with assessments at 1, 3, 6, 9, and 12 months Post-Permanent Device Activation.

Subjects who sign the informed consent will undergo evaluations to determine eligibility for the study based on the inclusion and exclusion criteria. Baseline assessments will also include measures for pain, disability, functioning, medication use, quality of life, depression and sleep.

Implantation and use of the Senza System will follow the Nevro Physician's Manual and supporting Manuals. Subjects will undergo a Trial Phase lasting up to 14 days to determine his/her response to SCS therapy. Following the Trial Phase with external device stimulation, subjects will be assessed for their pain, and those who have a successful Trial Phase will be eligible to proceed to permanent implantation of a SCS system.

Following permanent device implant, the IPG will be "activated" and thus, stimulation delivered on an ongoing basis for 12 months. At 1 month and 9 months following Post-Permanent Device Activation, assessments of pain and adverse events will be made. At 3, 6, and 12 months Post-Permanent Device Activation, subjects will be assessed for pain and adverse events as well as disability, functioning, medication use, quality of life, depression and sleep. Patient Global Impression of Change, Clinician Global Impression of Change and subject satisfaction will be recorded at 3 and 12 months Post-Permanent Device Activation.

ELIGIBILITY:
Inclusion Criteria:

1. Have been diagnosed with chronic, intractable pain of the upper limb and/or neck related to the cervical spine and/or neuropathic arm pain
2. Considering daily activity and rest, have average upper limb and/or neck pain intensity of ≥ 5 out of 10 cm on the Visual Analog Scale (VAS) at enrollment
3. Be an appropriate candidate for the surgical procedures required in this study based on the clinical judgment of the implanting physician
4. Be on stable pain medications, as determined by the Investigator, for at least 28 days prior to enrolling in this study and be willing to stay on those medications with no dose adjustments until activation of the permanently implanted SCS device
5. Be 18 years of age or older at the time of enrollment
6. Be willing and capable of giving informed consent
7. Be willing and able to comply with study-related requirements, procedures, and visits
8. Be capable of subjective evaluation, able to read and understand English-written questionnaires, and are able to read, understand and sign the written inform consent in English.
9. Have adequate cognitive ability to use a patient programmer and recharger as determined by the Investigator

Exclusion Criteria:

1. Have a medical condition or pain in other area(s), not intended to be treated with SCS, that could interfere with study procedures, as determined by the Investigator
2. Have evidence of an active disruptive psychological or psychiatric disorder as determined by a psychologist
3. Have a current diagnosis of a progressive neurological disease as determined by the Investigator
4. Have a current diagnosis of a coagulation disorder, bleeding diathesis, progressive peripheral vascular disease or uncontrolled diabetes mellitus
5. Have a condition that the Investigator determines would significantly increase perioperative risk
6. Significant cervical stenosis
7. Any previous history of surgery on the posterior elements (laminectomy, posterior fusion)
8. Be benefitting within from an interventional procedure and/or surgery to treat upper limb pain (Subjects should be enrolled at least 30 days from last benefit)
9. Have an existing drug pump and/or another active implantable device such as a pacemaker
10. Have a condition currently requiring or likely to require the use of MRI or diathermy
11. Have metastatic malignant disease or active local malignant disease
12. Have a life expectancy of less than 1 year
13. Have an active systemic or local infection
14. Be pregnant (if female and sexually active, subject must be using a reliable form of birth control, be surgically sterile or be at least 2 years post-menopausal)
15. Have within 6 months of enrollment a significant untreated addiction to dependency producing medications or have been a substance abuser (including alcohol and illicit drugs)
16. Be concomitantly participating in another clinical study
17. Be involved in an injury claim under current litigation -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects who respond to Senza SCS therapy (as assessed by VAS) for upper limb or neck pain | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Brad Gliner, Study Director — Nevro Corp
Locations (1):
- Nevro Corp., Redwood City, California, United States